CLINICAL TRIAL: NCT02610803
Title: Paroxysmal Atrial Fibrillation and Brief Runs of Premature Atrial Complexes in Patients With Acute Ischemic Stroke: A Historical Cohort Study
Brief Title: Paroxysmal Atrial Fibrillation in Patients With Acute Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Kristina Hoeg Vinther, Medical Doctor, Odense University Hospital
Other Study IDs: HISPACs
Record Dates: First submitted 2015-11-13; First posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Ischemic Stroke; Paroxysmal Atrial Fibrillation; Premature Atrial Complexes
Keywords: stroke; ischemic stroke; recurrent stroke; atrial fibrillation; premature atrial complexes; heart rhythm monitoring; cardiac telemetry
MeSH Terms: conditions — Ischemic Stroke; Atrial Fibrillation; Atrial Premature Complexes; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with ischemic stroke: Patients admitted with ischemic stroke from August 2008 to April 2011 (Retrospectively defined).

SUMMARY:
The purpose of this study is to estimate the clinical relevance of monitoring patients with acute ischemic stroke with 48 hours' inpatient cardiac telemetry in relation to evaluate the presence of brief runs of premature atrial complexes and new diagnosed atrial fibrillation. Furthermore to evaluate the prognostic significance of brief runs of premature atrial complexes in relation to develop atrial fibrillation, recurrent stroke/transient ischemic attack and death.

DETAILED DESCRIPTION:
Stroke is the second leading cause of death worldwide and it is well known that atrial fibrillation(AF) is a major risk factor for ischemic stroke. Paroxysmal AF can be difficult to detect because many cases are asymptomatic. In recent years prolonged cardiac rhythm monitoring of patients with ischemic stroke has showed an underestimated prevalence of AF. However, no optimal monitoring strategy is implemented in the clinic yet. This is the reason why research currently is focused on finding predictive risk markers of AF. Cohort studies of healthy individuals and stroke patients have shown that excessive premature atrial complexes (PACs) and brief runs of PACs are an emerging risk marker in helping to identifying patients in risk of having or developing AF. Despite this brief runs of PACs less than 30 s are today in everyday clinical practice perceived to be of no clinical significance.

The study population of ischemic stroke patients have all without known AF underwent ECG and 48 hours' inpatient cardiac telemetry as a clinical routine. In the medical record it is registered if patients had runs of PACs or new diagnosed AF.

All patients are registered in the Danish Stroke Registry, and all the baseline data on patients will be obtained from the registry.

The follow-up end August 2015 and information on AF, recurrent stroke and death will be obtained from medical records and the Funen Patient Administrative System, which is linked to the national Civil Registration System.

The purpose of this study is to estimate the clinical relevance of monitoring patients with acute ischemic stroke with 48 hours' inpatient cardiac telemetry in relation to evaluate the presence of brief runs of PACs and new diagnosed AF. Furthermore to evaluate the prognostic significance of brief runs of PACs in relation to develop AF and the prognostic significance of brief runs of PACs and AF in relation to recurrent stroke and death.

ELIGIBILITY:
Inclusion Criteria:

* admitted with ischemic stroke from August 2008-April 2011
* Registered in the Danish Stroke Registry

Exclusion Criteria:

* Hemorrhagic stroke
* No Danish civil registration
* no permanent address in Denmark during follow-up.
* patients with lack of telemetry data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke, admitted to our hospital between August 2008-April 2011
Sampling Method: Non-Probability Sample
Enrollment: 863 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Time to death or recurrent stroke | Up to 4 years

SECONDARY OUTCOMES:
Number of patients diagnosed with atrial fibrillation by 48 hours' continuous inpatient cardiac telemetry | up to 2 days
Number of patients diagnosed with runs of premature atrial complexes by 48 hours' continuous cardiac telemetry | up to 2 days
Time to develop atrial fibrillation in patients without know atrial fibrillation at admission. Registered in Medical journals and discharge letters. | Up to 4 years
Number of patients with atrial fibrillation having oral anticoagulant treatment at discharge. Data will be extracted from the Danish Stroke Registry. | to the day of discharge (up to 4 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Kristina H Vinther, MD, Principal Investigator
Locations (1):
- Department of Medical Research, OUH, Svendborg, Svendborg, Funen, Denmark